CLINICAL TRIAL: NCT04746586
Title: Identification and Characterization of Circulating microRNAs as Diagnostic Biomarkers in Adolescent Idiopathic Scoliosis
Brief Title: Identification of Circulating microRNAs in Adolescent Idiopathic Scoliosis
Acronym: IMIRSA
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: IDCE-AVEC 575-2020-Sper-IOR
Record Dates: First submitted 2020-11-26; First posted 2021-02-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Circulating microRNAs; Adolescent Idiopathic Scoliosis; Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma and circulating total RNA obtained from whole blood of enrolled AIS patients and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 20 patients with adolescent idiopathic scoliosis in a ratio of 5:1 between females and males will be enrolled.
  Interventions: Other: Circulating MiRNA indentification
- Controls: 10 healthy controls, of which 5 females and 5 males will be enrolled.
  Interventions: Other: Circulating MiRNA indentification

INTERVENTIONS:
Other: Circulating MiRNA indentification — Identification of circulating miRNA useful to discriminate between worsening and stable forms of AIS

SUMMARY:
The aim of the present study is to evaluate the expression of a large panel of microRNAs, already known and validated in other ortopedic pathologies and bone metabolism, in the plasma of Adolescent Idiopathic Scoliosis (AIS) patients. The deregulated microRNAs identified will be then validated and computational analyzes will determine their potential involvement in the metabolism of bone and/or cartilage tissue in order to correlate the results obtained with the clinical data of the AIS patients. The investigators aimed to develop a microRNAs panel to further validate in a larger population of AIS patients in order to produce a device for the diagnosis and prognosis of Molecular-based AIS.

DETAILED DESCRIPTION:
MATERIALS AND METHODS: 1) Collection of a venous blood sample from patients enrolled with AIS or controls, and subsequent separation of plasma; 2) Isolation of circulating total RNA from the plasma of AIS patients (Kit Invitrogen: Total RNA Isolation Reagent) and preparation of microRNA samples (TaqMan™ MicroRNA Reverse Transcription Kit); 3) Analysis of microRNA expression profiles by micro-array technique (Taqman Advanced miRNAs Human CardA + B); 4) Validation of deregulated microRNAs by single-qRT-PCR assay and computational functional analyses; and 5) In vitro studies to investigate the molecular role of the microRNAs identified within the mechanisms of bone remodeling.

Enrollment Procedures:

Patients considered eligible will be enrolled in the study, after providing a written informed consent. Healthy subjects (control group) will be recruited, on a voluntary basis, by means of an announcement published on the web page of the Rizzoli Orthopedic Institute (www.ior.it), "News" section.

Data Collection: Clinical data will be retrieved by patient's source document. A protocol-specific CRF reporting the results of the analyses will be provided. A CRF is required and should be completed for each included subject.

Ethics: The clinical trial protocol and its documents will be sent before initiating the study to the competent Authorities and Ethics Committees of each participating country for its approval. The responsible investigator will ensure that this study is conducted in agreement with either the most updated Declaration of Helsinki and all the international and local laws that apply to clinical trials and to patient protection. The protocol has been written, and the study will be conducted according to the principles of the ICH Harmonized Tripartite Guideline for Good Clinical Practice (ref: http://www.emea.eu.int/pdfs/human/ich/013595en.pdf).

Informed Consent: All patients will be informed, by the investigator, of the aims of the study, the possible risks and benefits that will derive from the study participation. The Investigator must clearly inform that the patient is free to refuse participation in the study and that can withdraw consent at any time and for any reason. The patients will be informed as to the strict confidentiality of their personal data, but the medical records of the patients enrolled may be reviewed for trial purposes by authorized individuals other than their treating physician. The informed consent procedure must conform to the ICH guidelines on Good Clinical Practice. This implies that "the written informed consent form should be signed and personally dated by the patient or by the patient's legally acceptable representative".

The Investigator must also sign the Informed Consent form, and will keep the original at the site and a copy of the original must be handed to the patient.

The competent ethics committee for each Institution participating to the study must validate local informed consent documents before the study can be opened. It will be emphasized that the participation is voluntary and that the patient is allowed to refuse further participation in the study whenever he/she wants. This will not prejudice the patient's subsequent care.

General Principles for Human Biological Material (HBM) collection: Human biological material (HBM) collection involves the collection and storage of biological material, residual biological material or derivatives in compliance with ethical and technical requirements. Biological material (blood samples) will be centralized and stored at Istituto Ortopedico Rizzoli - Dipartimento Rizzoli-Sicilia, Bagheria (Palermo). From here, the biological material will be used and stored according with the sample characteristic and applicable regulation.

Plasma and circulating total RNA obtained from blood will be stored inside sterile containers (falcon, tubes, eppendorf) in a freezer at the temperature of -80 °C at the Istituto Ortopedico Rizzoli - Dipartimento Rizzoli Sicilia.

The following principles apply to storage of HBM: (a) The Istituto Ortopedico Rizzoli will have a designated person responsible for collection and will act as a communication point; (b) The collected HBM should be documented, i.e. the amount remaining and its location. act as a communication point; and (c) The storage and use of biological material will take place in accordance with the standards of good laboratory practice (GLP) and applicable legislation.

Confidentiality: In order to ensure confidentiality of clinical trial data as disposed the national and European applicable regulation, data will be only accessible for the trial Sponsor and its designees, for monitoring/auditing procedures, the Investigator and collaborators, the Ethics Committee of each corresponding site and the Health Authority. Investigator and the Institution will allow access to data and source documentation for monitoring, auditing, Ethic Committee revision and inspections of Health Authority, but maintaining at all times subject personal data confidentiality as specified in the applicable regulation.

The Investigator must guarantee that patient anonymity is kept at all times and their identity must be protected from unauthorized persons and institutions.

All patients included in the study will be identified with a numeric code, so that no identifiable personal data will be collected. The Investigator must have and conserve a patients' inclusion registry where it figures the personal data of the patient: name, surname, address and corresponding identification code into the study, this register will be kept on the Investigator File.

Publication policy and data ownership: The principal investigator of the study is responsible for the final report, of the publication publish all the data collected as described in the protocol and will ensure that the data are reported responsibly and consistently. In particular, the publication of data deriving from the present study will take place independently of the results obtained. The transmission or dissemination of data, through scientific publications and / or presentation at conferences, congresses and seminars, will take place exclusively following the purely statistical processing of the same, or in an absolutely anonymous form. All the study data are owned by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Age between 11-17 years
* Diagnosis of idiopathic scoliosis with a Cobb angle> 10 °
* Minimum follow-up of two years
* Clinical data and radiological tests available and no surgical treatment prior to enrollment in the study

Controls:

* Age between 11-17 years
* Healthy subjects not affected by orthopedic and oncological diseases

Exclusion Criteria:

* Severe cognitive impairment or psychiatric disorders
* Patients with scoliosis due to secondary causes
* Women of childbearing age must not be pregnant

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A maximum number of 20 AIS patients in a ratio of 5:1 between females and males is expected to be enrolled; 10 healthy controls, of which 5 females and 5 males will be enrolled. Patients and control group (healthy volunteers) will be enrolled in the clinical trial only after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Isolation of circulating microRNAs from AIS patients and healthy controls | Within 24 hours of blood sampling
  Plasma samples will be obtained from blood samples of 20 AIS patients and 10 healthy subjects, collected in commercially available anticoagulant-treated tubes and centrifuged for 15 minutes at 2,000 x g. Circulating microRNAs will be isolated from the plasma samples by using commercially available miRNA Plasma Purification kit, specifically designed for purify high-quality microRNAs from plasma samples. Quantification and quality control of the purified circulating microRNAs will be determined through micro-spectrophotometry and microfluidics-based platforms.
Expression profiling of circulating microRNAs from AIS patients and healthy controls | Within 2 months of blood sampling
  The differentially expressed circulating microRNAs between AIS patients and healthy controls will be screened through micro-array technology using commercially available custom array microRNA cards, developed for profiling hundreds of unique human mature microRNAs known to be present in serum/plasma samples.

SECONDARY OUTCOMES:
Bioinformatics analysis of circulating microRNAs in AIS patients and healthy controls. | Within 3 months of blood sampling
  The analysis of microRNA profiling data will be carried out by considering the value of | log2 (HR) | ≥ 1.5 as differential expression limit of microRNA between the two groups of patients considered (AIS and control). The microRNAs not expressed in any sample will be excluded from the analysis.
  After data normalization, the differently expressed microRNAs will be analyzed with an analysis of hierarchical clusters. The TargetScan database (http://targetscan.org/) and the miRDB database (http://mirdb.org/miRDB/) will be used to predict the potential target genes of differentially expressed microRNAs.
  Target gene function analysis of differentially expressed miRNAs will be carried out on the Gene Ontology software (GO, http://meme.nbcr.net/meme/cgi-bin/gomo.cgi) and Kyoto Encyclopedia Genes and Genomes (KEGG, http: // www.genome .jp / kegg / expression)
Functional role of the circulating microRNAs related to AIS | Within 6 months of blood sampling
  To validate the microRNAs differentially expressed in the AIS patients compared to the healthy controls, specific qRT-PCR assays will be conducted in human bone cell lines (e.g. human primary osteoblasts, osteoclast, mesenchymal stem cells and chondrocyte cells). The role of microRNAs deregulated will be investigated in osteogenic, osteoclastic and chondrocyte differentiation by loss-of-function and gain-of-function experiments, in human bone cell lines (e.g. Runx2, ALP, Coll1A, OPN, OCN; TRAP, NFATc1, MMP9, CTSK; Coll2A, Sox9, ACAN). Viability assay (e.g. WST1 assay); apoptosis assay will be also performed (e.g. Annexin V staining assay, Caspase 3/7 assay and TUNEL detection methods).

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Toscano, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Dipartimento Rizzoli-Sicilia, Bagheria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Julien C, Gorman KF, Akoume MY, Moreau A. Towards a comprehensive diagnostic assay for scoliosis. Per Med. 2013 Jan;10(1):97-103. doi: 10.2217/pme.12.117. PMID 29783473
- [Result] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Result] Giampietro PF. Genetic aspects of congenital and idiopathic scoliosis. Scientifica (Cairo). 2012;2012:152365. doi: 10.6064/2012/152365. Epub 2012 Dec 31. PMID 24278672
- [Result] Asher MA, Burton DC. Adolescent idiopathic scoliosis: natural history and long term treatment effects. Scoliosis. 2006 Mar 31;1(1):2. doi: 10.1186/1748-7161-1-2. PMID 16759428
- [Result] Kaelin AJ. Adolescent idiopathic scoliosis: indications for bracing and conservative treatments. Ann Transl Med. 2020 Jan;8(2):28. doi: 10.21037/atm.2019.09.69. PMID 32055619
- [Result] Li Z, Yu X, Shen J. Environmental aspects of congenital scoliosis. Environ Sci Pollut Res Int. 2015 Apr;22(8):5751-5. doi: 10.1007/s11356-015-4144-0. Epub 2015 Jan 29. PMID 25628116
- [Result] Sparrow DB, Chapman G, Smith AJ, Mattar MZ, Major JA, O'Reilly VC, Saga Y, Zackai EH, Dormans JP, Alman BA, McGregor L, Kageyama R, Kusumi K, Dunwoodie SL. A mechanism for gene-environment interaction in the etiology of congenital scoliosis. Cell. 2012 Apr 13;149(2):295-306. doi: 10.1016/j.cell.2012.02.054. Epub 2012 Apr 5. PMID 22484060
- [Result] Li Z, Li X, Shen J, Zhang L, Chan MTV, Wu WKK. Emerging roles of non-coding RNAs in scoliosis. Cell Prolif. 2020 Feb;53(2):e12736. doi: 10.1111/cpr.12736. Epub 2019 Dec 12. PMID 31828859
- [Result] Chen C, Tan H, Bi J, Li Z, Rong T, Lin Y, Sun L, Li X, Shen J. Identification of Competing Endogenous RNA Regulatory Networks in Vitamin A Deficiency-Induced Congenital Scoliosis by Transcriptome Sequencing Analysis. Cell Physiol Biochem. 2018;48(5):2134-2146. doi: 10.1159/000492556. Epub 2018 Aug 15. PMID 30110682
- [Result] Garcia-Gimenez JL, Rubio-Belmar PA, Peiro-Chova L, Hervas D, Gonzalez-Rodriguez D, Ibanez-Cabellos JS, Bas-Hermida P, Mena-Molla S, Garcia-Lopez EM, Pallardo FV, Bas T. Circulating miRNAs as diagnostic biomarkers for adolescent idiopathic scoliosis. Sci Rep. 2018 Feb 8;8(1):2646. doi: 10.1038/s41598-018-21146-x. PMID 29422531